CLINICAL TRIAL: NCT04519944
Title: Edoxaban in Patients With Non-valvular Atrial Fibrillation Undergoing Percutaneous Coronary Intervention - German Non-interventional Study (ENCOURAGE-AF)
Brief Title: Edoxaban in Patients With Non-valvular Atrial Fibrillation Undergoing Percutaneous Coronary Intervention
Acronym: ENCOURAGE-AF
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Deutschland GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: DS-EDO-01-20-DE
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation; Antiplatelet therapy; Anticoagulation therapy; Percutaneous coronary intervention; Edoxaban
MeSH Terms: interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NVAF patients undergoing PCI: Patients with non-valvular atrial fibrillation (NVAF) who had successful percutaneous coronary intervention (PCI).
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — This is an observational, prospective study; no treatment will be administered.

SUMMARY:
This study is designed to gain real-world clinical data on the peri- and post-procedural usage of anticoagulation and antiplatelet therapy in patients with non-valvular atrial fibrillation (NVAF) undergoing successful percutaneous coronary intervention (PCI) treated with edoxaban.

DETAILED DESCRIPTION:
The study will assess real-world evidence data of anticoagulation and antiplatelet therapy in patients with NVAF undergoing PCI treated with edoxaban. The observation period will start 4 to 72 hours after removal of the guiding catheter of successful PCI in a hospital and ends 1 year after procedure. Follow-up telephone calls will take place approximately 1 month and 1 year after PCI. Real-world data of effectiveness of edoxaban and antiplatelet therapy, clinical events of interests, safety and quality of life (QoL) data of edoxaban will be collected.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Providing written informed consent (ICF) for participation in the study
* NVAF treated with edoxaban
* Successful PCI
* No planned elective cardiac intervention for the whole duration of the study (up to 1 year)
* Capability of patients for follow-up by telephone by the site for the whole duration of the study (up to 1 year)
* Availability of patients for follow-up by telephone by the site for the whole duration of the study (up to 1 year)
* Willingness of patients for follow-up by telephone by the site for the whole duration of the study (up to 1 year)
* Not simultaneously participating in any interventional study
* Life expectancy > 1 year

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will review database on 1200 participants with NVAF treated with Edoxaban in approximately 60 hospitals in Germany. All participants meeting the inclusion criteria and having given written informed consent will be enrolled. At least 25% of the participants should have acute coronary syndrome (ACS).
Sampling Method: Non-Probability Sample
Enrollment: 666 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Usage of Peri- and Post-procedural Anticoagulation and Antiplatelet Therapy in Patients With Non-valvular Atrial Fibrillation Undergoing Percutaneous Coronary Intervention | Up to 1 year follow up after PCI

SECONDARY OUTCOMES:
Number of Participants Reporting Clinical Events of Interest in Patients With Non-valvular Atrial Fibrillation Undergoing Percutaneous Coronary Intervention | Up to 1 year follow up after PCI
  Bleeding (major, minor, CRNM), stroke, myocardial infarction (MI), percutaneous coronary intervention (PCI), and death will be assessed.
EQ-5D-5L Assessment in Patients With Non-valvular Atrial Fibrillation Undergoing Percutaneous Coronary Intervention | Up to 1 year follow up after PCI
Number of Hospital Admissions in Patients With Non-valvular Atrial Fibrillation Undergoing Percutaneous Coronary Intervention | Up to 1 year follow up after PCI
Duration of Hospital Admission in Patients With Non-valvular Atrial Fibrillation Undergoing Percutaneous Coronary Intervention | Up to 1 year follow up after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (66):
- Germany (66):
  - Zentralklinik Bad Berka, Bad Berka
  - SLK-Kliniken Heilbronn GmbH Klinikum am Plattenwald, Bad Friedrichshall
  - Kerckhoff-Klinik GmbH, Bad Nauheim
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Schüchtermann-Schiller'sche Kliniken Bad Rothenfelde GmbH & Co. KG, Bad Rothenfelde
  - Charité - Campus Mitte, Berlin
  - Charité - Campus Benjamin Franklin, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - GFO-Kliniken, Standort St.-Marienhospital Bonn, Bonn
  - StädtischesKlinikum Brandenburg, Brandenburg
  - Klinikum Braunschweig, Braunschweig
  - Klinikum Chemnitz, Chemnitz
  - REGIOMED-KLINIKEN GmbH, Klinikum Coburg, Coburg
  - Krankenhaus der Augustinerinnen Köln, Cologne
  - St. Vinzenz-Hospital Köln, Cologne
  - Universitätsklinikum Köln, Cologne
  - Evangelisches Krankenhaus Kalk gGmbH, Cologne
  - Kreiskrankenhaus Demmin GmbH, Demmin
  - Klinikum Lippe Detmold, Detmold
  - St. Johannes-Hospital Dortmund, Dortmund
  - Herzzentrum Dresden GmbH Universitätsklinik an der Technischen Universität Dresden, Dresden
  - Krankenhaus Eggenfelden, Eggenfelden
  - Universitätsklinikum Essen, Essen
  - CCB Cardioangiologisches Centrum Bethanien, Frankfurt
  - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main
  - Universitäts Herzzentrum Freiburg Bad Krozingen, Freiburg im Breisgau
  - Klinikum Fürth, Fürth
  - SRH Wald-Klinikum Gera, Gera
  - Universitätsklinikum Greifswald, Greifswald
  - Klinikum Gütersloh, Gütersloh
  - Asklepios Klinik St. Georg, Hamburg
  - Asklepios Kliniken Hamburg GmbH - Aklepios Klinik Barmbek, Hamburg
  - Asklepios Klinikum Harburg, Harburg
  - SLK-Kliniken Heilbronn, Heilbronn
  - Klinikum Nordfriesland, Husum
  - Universitätsklinikum Jena, Jena
  - SRH Klinikum Karlsbad-Langensteinbach GmbH, Karlsbad
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Gemeinschaftsklinikum Mittelrhein gGmbH, Ev. Stift St. Martin, Koblenz
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - UKSH Lübeck, Lübeck
  - Klinikum Lüdenscheid, Märkische Gesundheitsholding GmbH & Co. KG, Lüdenscheid
  - Carl-von-Basedow-Klinik Saalekreis GmbH, Merseburg
  - Technische Universität München, Klinikum rechts der Isar, München
  - München Klinik gGmbH, Klinik Neuperlach, München
  - St. Franziskus-Hospital GmbH, Münster
  - Klinikum Oldenburg AöR, Universitätsklinik für Innere Medizin - Kardiologie, Oldenburg
  - St. Vincenz Krankenhaus, Paderborn
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Quedlinburg
  - Universitätsmedizin Rostock, Rostock
  - Herz-Kreislauf-Zentrum Rotenburg, Rotenburg an der Fulda
  - Leopoldina, Schweinfurt
  - Klinikum Westmünsterland GmbH, Stadtlohn
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
  - SRH Zentralklinikum Suhl, Innere Medizin I, Suhl
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Herzzentrum Saar, Völklingen
  - Kliniken Nordoberpfalz AG, Weiden
  - GRN-Klinik Weinheim, Weinheim
  - Klinikum Wilhelmshaven gGmbH, Wilhelmshaven
  - Petrus-Krankenhaus Wuppertal, Wuppertal
  - Universitätsklinikum Würzburg, Würzburg
  - Heinrich-Braun-Klinikum Zwickau, Zwickau

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Baldus S, Beyer-Westendorf J, Mollmann H, Rottbauer W, Beyerlein E, Goette A. Edoxaban in patients with non-valvular atrial fibrillation after percutaneous coronary intervention: ENCOURAGE-AF design. Sci Rep. 2023 Oct 25;13(1):18215. doi: 10.1038/s41598-023-44345-7. PMID 37880316